CLINICAL TRIAL: NCT03087058
Title: A Phase 2, Open-Label, Multiple Dose Study to Evaluate the Pharmacodynamic Effects, Safety, and Tolerability of Patiromer for Oral Suspension in Children and Adolescents 2 to < 18 Years of Age With Chronic Kidney Disease and Hyperkalemia
Brief Title: Pharmacodynamic & Safety of Patiromer in Children & Adolescents (2-<18 Yrs) With Chronic Kidney Disease and Hyperkalemia
Acronym: EMERALD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on 13 May 2022 due to a modification to the PIP/PSP
Sponsor: Vifor Pharma, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RLY5016-206p; 2016-002785-31 (EudraCT Number)
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Results first posted 2022-09-26 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Hyperkalemia
Keywords: Treatment of Hyperkalemia; Hyperkalemia; Potassium; Chronic Kidney Disease
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic | interventions — patiromer; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Patiromer for age 12 to < 18 years
  Interventions: Drug: Patiromer
- Cohort 2 (Experimental): Patiromer for age 6 to < 12 years
  Interventions: Drug: Patiromer
- Cohort 3 (Experimental): Patiromer for age 2 to < 6 years
  Interventions: Drug: Patiromer

INTERVENTIONS:
Drug: Patiromer — 4.2 g/day, 8.4 g/day and 16.8 g/day
  Other Names: Veltassa; RLY5016 for Oral Suspension
  Arms: Cohort 1
Drug: Patiromer — 2 g/day, 4 g/day and 8 g/day
  Other Names: Veltassa; RLY5016 for Oral Suspension
  Arms: Cohort 2
Drug: Patiromer — 1 g/day, 2 g/day and 4 g/day
  Other Names: Veltassa; RLY5016 for Oral Suspension
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to evaluate the change in serum potassium levels from start of treatment to Day 14, when patiromer is administered at different doses, once daily, in children 2 - < 18 years of age with chronic kidney disease (CKD) and hyperkalemia (too much potassium in the blood). Another purpose of the study is to evaluate the safety and tolerability of patiromer in children 2 - < 18 years of age with CKD and hyperkalemia.

DETAILED DESCRIPTION:
Up to 54 subjects, 2 - < 18 years of age with CKD (estimated glomerular filtration rate [eGFR] < 90 mL/min/1.73 m2 ) and hyperkalemia (two potassium measurements of 5.1 to < 6.5 mEq/L performed on separate days) will be enrolled in this open-label, multiple-dose, Phase 2 study.

The study will include two treatment phases: Pharmacodynamic (PD; drug effect on potassium) / Dose Finding Phase consisting of the initial 14-day dose finding period followed by an up to 5.5-month Long-Term Treatment Phase for a total study participation duration for individual subjects of up to 6.5 months (includes a 2 week follow up period).

ELIGIBILITY:
Inclusion Criteria:

* Written assent (when applicable) and written informed consent by a legally authorized representative provided prior to participation in the study
* Age 2 - <18 years old
* CKD defined by the estimated glomerular filtration rate (eGFR) <90 mL/min/1.73m2, including renal transplant subjects, based on local creatinine measurement at screening
* Two potassium measurements of 5.1 to < 6.5 mEq/L performed on separate days
* In the opinion of the study doctor, is expected to require treatment for hyperkalemia for at least 6 month
* If taking any renin-angiotensin-aldosterone system inhibitors (RAASi) beta blockers or diuretic medications, must be on a stable dose for at least 28 days prior to Screening
* Negative pregnancy test in females of child-bearing potential

Exclusion Criteria:

* Pseudohyperkalemia due to hemolysis or to abnormally high numbers of platelets (>500,000/mm3), leukocytes (>70,000/mm3), or erythrocytes (hematocrit >55%) at Screening based on results obtained locally
* Evidence of potassium-related electrocardiogram (ECG) changes at Screening
* Any of the following kidney conditions: maintenance hemodialysis or peritoneal dialysis, renal artery stenosis, and acute kidney injury or a history of acute renal insufficiency in the past 3 months
* Severe disorder of stomach or intestines including surgery that could affect gastrointestinal transit of the drug
* Increased liver enzymes (ALT, AST > 3 times upper limit of normal) at Screening
* Active cancer, currently on cancer treatment or history of cancer in the past 2 years (except for non-melanoma skin cancer)
* Heart or liver transplant, or anticipated need for transplant during the study treatment period including a scheduled kidney transplant recipient. (Note: patients currently on a kidney transplant wait list are not excluded unless there is an identified donor).
* Alcohol abuse or substance use disorder within 1 year of Screening
* Subjects currently being treated with or having taken any one of the following medications (includes resins) in the 7 days prior to Screening: sodium or calcium polystyrene sulfonate, drospirenone
* Use of certain medications that can affect blood potassium levels if doses have not been stable for at least 14 days prior to Screening or if doses are anticipated to change during the 14-day PD / Dose Finding Phase
* Use of investigational product within 30 days of screening or within 5 half-lives, whichever is longer
* Known hypersensitivity to patiromer or its components
* In the opinion of the Investigator, any medical condition, uncontrolled systemic disease, or serious intercurrent illness that would significantly decrease study compliance or jeopardize the safety of the subject or potentially affect the quality of the data

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Platon, MD, PhD, Study Director — Vifor Pharma, Inc.
Locations (30):
- United States (10):
  - Investigator Site 1107, Palo Alto, California
  - Investigator Site 1101, Kansas City, Kansas
  - Investigator Site 1103, Baltimore, Maryland
  - Investigator Site 1102, The Bronx, New York
  - Investigator Site 1105, Cincinnati, Ohio
  - Investigator Site 1108, Pittsburgh, Pennsylvania
  - Investigator Site 1104, Amarillo, Texas
  - Investigator Site 1109, Dallas, Texas
  - Investigator Site 1113, Houston, Texas
  - Investigator Site 1106, Madison, Wisconsin
- Investigator Site 1401, Sofia, Bulgaria
- Investigator Site 1902, Vancouver, British Columbia, Canada
- Georgia (5):
  - Investigator Site 3915, Tbilisi
  - Investigator Site 3913, Tbilisi
  - Investigator Site 3911, Tbilisi
  - Investigator Site 3912, Tbilisi
  - Investigator Site 3914, Tbilisi
- Germany (4):
  - Investiagor Site 4314, Cologne
  - Investigator Site 4312, Essen
  - Investigator Site 4313, Hanover
  - Investigator Site 4311, Heidelberg
- Poland (6):
  - Investigator Site 5401, Bialystok
  - Investigator Site 5404, Gdansk
  - Investigator Site 5406, Krakow
  - Investigator Site 5402, Lodz
  - Investigator Site 5403, Lublin
  - Investigator Site 5405, Warsaw
- Ukraine (3):
  - Investigator Site 7906, Dnipro
  - Investigator Site 7903, Kharkiv
  - Investigator Site 7904, Kyiv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Patiromer administrated to pediatric participants (12 to <18 years of age), with chronic kidney disease (CKD) and hyperkalemia.
  The starting dose levels of Patiromer for Cohort 1 were: 4.2 g/day, 8.4 g/day and 16.8 g/day, starting with the lowest dose level, depending on the participant's median weights.
  Once-daily administration up to 26 weeks including screening at Day 1 followed by 14-days (Pharmacodynamic dose-finding phase), 22 weeks (Long-term treatment phase), and a 2-week follow-up period consisting of 1 follow-up visit and 1 follow-up phone call.
- Cohort 2: Patiromer administrated to pediatric participants (6 to <12 years of age), with chronic kidney disease (CKD) and hyperkalemia.
  The starting dose levels of Patiromer for Cohort 2 were: 2 g/day, 4 g/day and 8 g/day, starting with the lowest dose level, depending on the participant's median weights.
  Once-daily administration up to 26 weeks including screening at Day 1 followed by 14-days (Pharmacodynamic dose-finding phase), 22 weeks (Long-term treatment phase), and a 2-week follow-up period consisting of 1 follow-up visit and 1 follow-up phone call.
- Cohort 3: Patiromer was planned to be administrated to pediatric participants (2 to <6 years of age), with chronic kidney disease (CKD) and hyperkalemia. However, the trial was terminated by sponsor decision on the 13 July 2022. The PD effects, safety and tolerability of patiromer in the population aged from 0 to <6 will be assessed in a new trial with the protocol number RLY5016-208p.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 14 | 9 | 0 (Vifor believes the 23 enrolled subjects in Cohort 1 and 2 are representative of patients with hyperkalaemia due to CKD 6 to <18 years of age and that data are sufficient to support assessment of the PD effects, safety, and tolerability of patiromer in this population. The trial was terminated by sponsor decision on the 13 July 2022. The PD and safety of patiromer in the population aged from 0 to <6 will be assessed in a new trial with the protocol number RLY5016-208p.)
Completed | 12 | 9 | 0
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2: Patiromer administrated to pediatric participants (6 to <12 years of age), with chronic kidney disease (CKD) and hyperkalemia.
  The starting dose levels of Patiromer for Cohoer1 1 were: 2 g/day, 4 g/day and 8 g/day, starting with the lowest dose level, depending on the participant's median weights.
  Once-daily administration up to 26 weeks including screening at Day 1 followed by 14-days (Pharmacodynamic dose-finding phase), 22 weeks (Long-term treatment phase), and a 2-week follow-up period consisting of 1 follow-up visit and 1 follow-up phone call.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 9 | 23
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.99) | 8.0 (2.00) | 12.0 (3.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 11 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 0 | 2
  Ukraine | 6 | 7 | 13
  Poland | 1 | 1 | 2
  Georgia | 3 | 1 | 4
  Germany | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Potassium Levels
Time Frame: from Baseline to Day 14
Population: The efficacy population includes all subjects who have taken at least 1 dose of patiromer.
  As the safety population and efficacy population are the same in this study, all analyses are displayed with 1 population.
Measure: Mean (Standard Deviation); unit: mEq/l
Groups:
- Cohort 2: Patiromer administrated to pediatric participants (6 to < 12 years of age), with chronic kidney disease (CKD) and hyperkalemia.
  The starting dose levels of Patiromer for Cohoer1 1 were: 2 g/day, 4 g/day and 8 g/day, starting with the lowest dose level, depending on the participant's median weights.
  Once-daily administration up to 26 weeks including screening at Day 1 followed by 14-days (Pharmacodynamic dose-finding phase), 22 weeks (Long-term treatment phase), and a 2-week follow-up period consisting of 1 follow-up visit and 1 follow-up phone call.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 14 | 9
mEq/l | -0.50 (0.542) | -0.14 (0.553)

2. Secondary Outcome: Proportion of Subjects With Serum Potassium Levels in the Range of 3.8 - 5.0 mEq/L
Description: Day 14: Initial PD / Dose Finding Phase. Week 26: Long-Term Treatment Phase.
Time Frame: Day 14 and Week 26
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants (%)
Groups:
- Cohort 1: Patiromer administrated to pediatric participants (12 to < 18 years of age), with chronic kidney disease (CKD) and hyperkalemia.
  The starting dose levels of Patiromer for Cohort 1 were: 4.2 g/day, 8.4 g/day and 16.8 g/day, starting with the lowest dose level, depending on the participant's median weights.
  Once-daily administration up to 26 weeks including screening at Day 1 followed by 14-days (Pharmacodynamic dose-finding phase), 22 weeks (Long-term treatment phase), and a 2-week follow-up period consisting of 1 follow-up visit and 1 follow-up phone call.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 14 | 9
percentage of participants (%)
  Day 14 | 50.0 [23.0 to 77.0] | 12.5 [0.3 to 52.7]
  Week 26 | 81.8 [48.2 to 97.7] | 22.2 [2.8 to 60.0]

ADVERSE EVENTS:
Time Frame: During treatment period up to 26 weeks after randomization.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/9
Other Adverse Events (participants affected / at risk) | 10/14 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=14) | Cohort 2 (N=9)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Human herpesvirus 6 infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Urine output increased (Investigations) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Dysphoria (Psychiatric disorders) | 1 (1) | 0 (0)
Psychomotor retardation (Psychiatric disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT03087058/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT03087058/SAP_001.pdf